CLINICAL TRIAL: NCT00330122
Title: Restoration of the Radial Length in Compound Wrist Fractures Using Anterior Locking Plates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC-05-01; 2005/20 (CCPPRB); 2006/0017 (DGS)
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2006-05-25 (Estimated); Status verified 2006-05

CONDITIONS: Articular Displaced Fractures of the Lower End of the Radius
Keywords: radius articular displaced fractures; fore locked plate; external radiocarpal fixer

INTERVENTIONS:
Procedure: fore locked plate
Procedure: external radiocarpal fixer

SUMMARY:
The fractures of the wrist, affecting the distal end of the radius are frequent, in particular in the old subject and/or osteoporotic. Beside the simple fractures treated by mini-invasive surgical methods, there is a considerable number of strong comminuted fractures for which no method of osteosynthesis proves completely satisfactory, especially on osteoporotic bone. However, the restitution of the anatomy remains the principal concern of the surgeon eager to ensure a good functional result to its patient, with the proviso that the least aggressive possible method is used.

Until now, it is of use to rather largely use the external fixer bridging the radiocarpal articulation to maintain the length of the radius, more or less associated with an another method of internal osteosynthesis with minima. The major disadvantage of this kind of assembly is the high rate of neuroalgodystrophic syndromes of the wrist and losses of reduction, sometimes generators of painful after-effects and serious stiffening. These after-effects which are sometimes definitive can be very disabling when they occur among active people, a fortiori when they touch the dominant side.

The recent alternative to the use of the external fixer is the use of the plates with locking screws, affixed on the foreface of the radius, maintaining the length of the radius but not bridging the articulation. Thus, this kind of osteosynthesis does not generate ligamentary distraction nor of the radiocarpal capsule, factors which would be prevalent in the release of the algodystrophy and of the stiffening. On the other hand, this method of osteosynthesis is more invasive than the installation of an external fixer, because it requires the access of the foreface of the radius and cannot be practised in a percutaneous way. At present, there is any randomized comparative study, the published studies being only comparative retrospective and not controlled, carried out on nonhomogeneous series of fractures.

The principal objective of our study is to evaluate the interest of the locking plates in the maintenance of the radial length in the comminuted fractures of the distal end of the radius.

It is about a prospective, multicentric, randomized study in 2 parallel groups carried out patients from 40 to 80 years hospitalized in a service of Osseous Surgery.

Patients: articular displaced fractures of the lower end of the radius with strong metaphysar comminution (groups M3 and M4 of the classification MEC) with an important shortening of the radius, measured by a radio-ulnar index higher than 4 mm compared to the opposite side. Are excluded the articular explosions type E4. The patients of more than 40 years, autonomous and active, able to give an assent for the participation in a clinical study are included.

Treatment. The first group of patients would be treated by fore locked plate possibly associated with pins. The immobilization would be limited to a antibrachiopalmar splint for 45 days. If, peroperatively, a sufficient stability of the fracture cannot be obtained by the plate alone, and that a complementary stabilization by fixer proves to be necessary, then the case will be entered like a failure of stabilization by locked plate.

The second group of patients would be treated by external radiocarpal fixer in neutralization possibly associated with an internal osteosynthesis with minima (percutaneous pins). The fixer would be left in place during 45 days.

The reeducation would consist in the 2 groups of an active mobilization of the fingers at the beginning, then of an active reeducation of the wrist in flexion/extension and pronosupination starting from the 45th day.

About fifty patients should be included in each group, with a collection of the clinical and radiographic results at 21 days, 45 days, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* articular displaced fractures of the lower end of the radius with strong metaphysar comminution (groups M3 and M4 of the classification MEC) with an important shortening of the radius, measured by a radio-ulnar index higher than 4 mm compared to the opposite side
* age < 40 years
* autonomous and active
* able to give an assent for the participation in a clinical study

Exclusion Criteria:

* articular explosions type E4

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-03; Study Completion 2006-05

PRIMARY OUTCOMES:
maintenance of the radial length 3 month after surgery

SECONDARY OUTCOMES:
maintenance of the radial length 6 month after surgery
complication and algodystrophia after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MASSIN, Professor, Study Director — UH of Angers
Locations (3):
- France (3):
  - UH of Angers, Angers
  - UH of Besancon, Besançon
  - UH of Tours, Tours